CLINICAL TRIAL: NCT05206240
Title: Efficacy of Extracorporeal Shock Wave Therapy and Assessment Strategy Through a Novel Gait Analysis Tool for Post-stroke Spasticity During COVID-19 Pandemic
Brief Title: Extracorporeal Shock Wave Therapy and Assessment Strategy Through a Novel Gait Analysis Tool for Post-stroke Spasticity
Status: Completed | Type: Observational
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Emanuela Elena Mihai, Principal Investigator, Carol Davila University of Medicine and Pharmacy
Other Study IDs: 2090
Record Dates: First submitted 2021-12-24; First posted 2022-01-25 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Stroke, Ischemic; Stroke Hemorrhagic; Spasticity, Muscle; Spastic Gait
Keywords: stroke; spasticity; neurological rehabilitation; radial extracorporeal shock wave therapy; gait analysis system
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke; Muscle Spasticity; Gait Disorders, Neurologic; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: The patients considered eligible will form the study group and will start the conventional physical therapy program and radial extracorporeal shock wave therapy delivery (rESWT).
  Interventions: Other: Radial extracorporeal shock wave therapy and conventional physical therapy

INTERVENTIONS:
Other: Radial extracorporeal shock wave therapy and conventional physical therapy — The conventional physical therapy program will consist of verticalization strategies, range of motion exercises, muscle stretching and strengthening exercises, stance and balance training, core stability exercises, gait training, functional training, cryotherapy or local heat for 1h/day, 5 days/week for 2 weeks.
  Regarding the rESWT delivery, 2000 shots will be applied on the triceps surae myotendinous junction with a frequency of 10 Hz and an energy density of 60 mJ, 7 min/session, 1 session/week for 2 weeks.

SUMMARY:
The aim of this study is to objectively evaluate the effectiveness of radial extracorporeal shock wave therapy (rESWT) and conventional physical therapy program on the gait pattern through a new gait analysis system which encompasses spatiotemporal and kinematic parameters and to correlate the findings with the clinical evaluation.

DETAILED DESCRIPTION:
The aim of this observational study was to objectively evaluate the effects of radial extracorporeal shock wave therapy and conventional physical therapy program on the gait pattern, spatiotemporal variables (step length, step cycle time, stance foot flexion-extension, foot stance pronation-supination, and foot swing flexion-extension), and kinematic parameters (trunk flexion-extension, trunk lateral flexion, hip flexion-extension, knee flexion-extension, ankle flexion-extension) through a new gait analysis system and correlate the findings with clinical outcomes such as Modified Ashworth scale (MAS), passive range of motion (PROM), Clonus score, Visual Analogue Scale (VAS), Tinetti Assessment Tool, Functional Ambulation Categories (FAC).

The gait pattern of post-stroke patients before and after rESWT delivery and conventional rehabilitation program will be assessed clinically and also through an instrumented treadmill (Walker View) in terms of spatiotemporal and kinematic gait parameters.

ELIGIBILITY:
Inclusion Criteria:

* suffered from a hemorrhagic or ischemic stroke and they were in the subacute or chronic phase;
* had no history of previous stroke;
* had lower limb post- stroke spasticity and spasticity grade ≥1 on the Modified Ashworth Scale (MAS);
* pain intensity measured on Visual Analogue Scale (VAS) ≥1;
* ability to stand and walk unassisted for at least 30 seconds;
* adult patients (>18 years old).

Exclusion Criteria:

* other neurological, musculoskeletal, orthopaedic, or cardiovascular conditions; -- severe cognitive impairment, severe aphasia or inability to understand or execute instructions;
* changes in antispastic medication and dose or changes in the analgesic medication;
* myopathy;
* severe spasticity grade;
* visual field disorders or hemineglect;
* anticoagulants or any contraindication to receive radial extracorporeal shock wave therapy (rESWT), or any contraindication to receive physical therapy sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients from the Physical and Rehabilitation Medicine Department stating the eligibility criteria
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Spasticity grade change | Change from baseline Modified Ashworth Scale at 14 days
  Modified Ashworth Scale (MAS); ranges from 0 (no increase in muscle tone) to 5 (rigid limb in flexion or extension). The lower the score, the lower spasticity grade, thus a better outcome.

SECONDARY OUTCOMES:
Ankle passive range of motion change | Change from baseline Passive Range of Motion at 14 days
  Passive range of motion (PROM); flexion 0-30 degrees, extension 0-50 degrees, pronation 0-30 degrees, supination 0-60 degrees. Higher scores define augmented, better range of motion.
Pain intensity change | Change from baseline Visual Analogue Scale at 14 days
  Visual Analogue Scale (VAS); the greater the value on the 0.1 meters line, the greater the pain intensity starting from 0 (no pain at all) to 10 (the highest pain intensity ever experienced).
Step length change | Change from baseline step length at 14 days
  Step length (meters); ranges from 0-0.5 meters, the higher the step length leads to better outcome.
Knee flexion-extension change | Change from baseline knee flexion-extension at 14 days
  Knee flexion-extension; Maximum and minimum angle value in the sagittal plane of knee, from 0 degrees in full extension to 140-150 degrees in maximum flexion.

CONTACTS AND LOCATIONS:
Overall Officials: Mihai Berteanu, Study Director — Elias University Emergency Hospital, Bucharest, Romania
Locations (1):
- Elias University Emergency Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No